CLINICAL TRIAL: NCT05969184
Title: Palbociclib Combine With Endocrine Therapy and Anti-HER2 Therapy in HR Positive and HER2 Positive Advanced Breast Cancer
Brief Title: Palbociclib Combine With Anti-HER2 Therapy in Triple Positive ABC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Li Huiping, Head of the department of breast oncology, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABC015
Record Dates: First submitted 2022-12-14; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — pertuzumab

STUDY DESIGN:
Masking Description: we have only one single center participant and none of the roles in research needed to be mask
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- four-drug treatment group (Experimental): CDK4/6 inhibitor (Qilu): 125mg, oral Qd from the 1st to the 21st day of the 28 day cycle Trastuzumab (Hanquyou): on the first day of the 21 day cycle, the initial dose was 8mg/kg, and the intravenous infusion was 90 minutes; Every 3 weeks thereafter, the dose is 6mg/kg, and the intravenous infusion is 30~90 minutes Pertuzumab: on the first day of the 21 day cycle, the initial dose was 840mg, intravenous infusion was 60 minutes, and then once every 3 weeks, the dose was 420mg, and the infusion time was 30-60 minutes.
  Letrozole selected by the doctor: 2.5mg, oral Q24H or exemestane from the 1st to the 21st day of the 21 day cycle: 25mg, oral Q24H from the 1st to the 21st day of the 21 day cycle. The efficacy is evaluated every 2 months (CR, PR, SD, PD).
  Interventions: Drug: CDK4/6 inhibitor (Qilu),Trastuzumab (Hanquyou)

INTERVENTIONS:
Drug: CDK4/6 inhibitor (Qilu),Trastuzumab (Hanquyou) — CDK4/6 inhibitor (Qilu) have got the cFDA approval and Trastuzumab (Hanquyou) have few data on combination use, this two drugs need clinical treatment data
  Other Names: Pertuzumab,Letrozole,exemestane

SUMMARY:
This study is to find out that if HER-2 positive and HR positive patients could benefit from trastuzumab and pertuzumab combined with palbociclib and endocrine therapy.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, multicenter, phase II clinical study. Subjects were eligible for screening and entered the trial period after enrollment and received treatment with palbociclib（125mg/day), trastuzumab(8 mg→6mg/every 3 week), pertuzumab(840 mg→420mg/every 3 week), combined with endocrine therapy until disease progression, or intolerable toxicity, or withdrawal of informed consent, or discontinuation of medication at the investigator 's discretion. On-study imaging assessments were performed according to RECIST 1.1 criteria and the site assessment was final.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form and agree to comply with the requirements of the research protocol
* Recurrent or metastatic breast cancer confirmed by histology or cytology that cannot be operated, and has not received systematic treatment for recurrent or metastatic breast cancer.
* Estrogen receptor ER is positive (positive staining of ≥ 1% of tumor cell nucleus is positive) and HER2 is positive (immunohistochemistry is 3+, and/or 2+, and ISH is positive)
* Age ≥ 18 years old.
* ECOG physical status score is 0-1.
* Life expectancy ≥ 3 months.
* Be in a postmenopausal state.
* Suffer from one of the following diseases defined in RECIST 1.1, and the target lesion is not suitable for surgical treatment; The target lesion has not received radiotherapy or relapses in the radiotherapy field:

  * At least one measurable lesion as the target lesion confirmed by CT or MRI
  * Non measurable disease with only bone metastasis (osteogenic disease, osteolytic disease or osteolytic osteogenic mixture)
* Appropriate hematopoietic function, liver function and kidney function

Exclusion Criteria:

* Visceral crisis, severe organ dysfunction accompanied by clinical symptoms and signs, and the clinician judges that it is necessary to receive chemotherapy based treatment as soon as possible to obtain disease relief, including but not limited to the following situations: liver metastasis accompanied by a rapid increase of more than 1.5 times of bilirubin or more than 3 times of transaminase; Or pulmonary metastasis with dyspnea at rest; Carcinomatous lymphangitis; Bone marrow metastasis was accompanied by severe decrease of hematopoietic function; As well as asthma, inflammatory breast cancer, etc.
* The subject has cancerous meningitis or has untreated central nervous system metastasis; Those who have received systematic and radical brain metastasis treatment (radiotherapy or surgery) in the past, and have been stable for at least 1 month as confirmed by imaging, and have stopped systemic hormone treatment (dose>10mg/day prednisone or other effective hormones) for more than 2 weeks, and have no clinical symptoms can be included.
* over 2 kind of Systematic treatment for metastatic breast cancer, including chemotherapy, endocrine therapy and biological targeting therapy, has been used previously.
* Have received any treatment of CDK4 and CDK6 inhibitors (or participated in any clinical trial of CDK4 and CDK6 inhibitors that have not been exposed).
* Have received radiotherapy within 28 days before enrollment. It is allowed to receive radiotherapy for relieving metastatic bone pain before enrollment, but the irradiated medullary bone shall not exceed 30% of the total amount.
* Patients with uncontrolled lung disease, severe infection, active digestive tract ulcer requiring treatment, coagulation disorders, severe uncontrolled diabetes, connective tissue disease or bone marrow function depression and other diseases cannot tolerate the study drug treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 2 year
  calculated from the first administration time of the study drug to the disease progress or death. If the patient does not have PD or death on the study deadline, or has received other anti-tumor treatment, the deadline shall be the last efficacy evaluation result before the deadline or the start date of other anti-tumor treatment (whichever occurs first)

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 year
  it refers to the proportion of patients who have the best response effect of CR or PR from the beginning of receiving the treatment plan of this study to the time when the patient's disease progresses out of the group. Tumor imaging examination shall be performed at baseline and every 2 cycles (6 weeks) thereafter. If the patient reaches CR or PR, it shall be confirmed after 6 weeks. If patients delay treatment due to toxicity, they still need to receive efficacy evaluation every 6 weeks.
Disease control rate (DCR) | 2 year
  refers to the proportion of patients who have achieved complete remission (CR), partial remission (PR) or stable disease (SD) at least once after receiving the treatment of this study protocol
Duration of remission (DoR) | 2 year
  from the date when CR or PR evidence was first found to the date when objective progress occurred or the date of death due to any reason, whichever is earlier. If the patient does not know whether the patient is PD or dead at the deadline of the study, the date of the last complete objective progression free disease assessment shall be taken as the data deletion.
Total survival (OS) | 2 year
  calculated from the first administration of the study drug to the death due to any reason.The OS of patients who still survived at the last follow-up is counted as the data deletion based on the time of the last follow-up. For patients who lost the interview, their OS was counted as data deletion based on the last confirmed survival time before the lost interview. The OS of data deletion is defined as the time from grouping to deletion
time to treatment failure(TTF) | 2 year
  calculated from enrolled in the study to stop treatment resulted in any reason

CONTACTS AND LOCATIONS:
Overall Officials: Yaxin Liu, Dr, Study Chair — Peking University Cancer Hospital and Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Yaxin Liu, Beijing, None Selected

IPD SHARING:
Plan to Share IPD: No
research plan would be share after completion of patients enroment.